CLINICAL TRIAL: NCT05622799
Title: Mind-Body Medicine Training for Incarcerated Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Mind-Body Medicine (Other)
Collaborators: Simon Family Foundation (Unknown)
Responsible Party: Principal Investigator, Julie K. Staples, Research Director, The Center for Mind-Body Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CMBMIndianaPrison001
Record Dates: First submitted 2022-11-07; First posted 2022-11-21 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Resilience
Keywords: Mind-body therapies; Resilience; Prisoners; Meditation

STUDY DESIGN:
Intervention Model Description: Non-controlled repeated measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mind-Body MedicineTraining (Experimental): A two part (4 days for each part) mind-body medicine training program
  Interventions: Behavioral: Mind-Body Medicine Training Program

INTERVENTIONS:
Behavioral: Mind-Body Medicine Training Program — A mind-body medicine training program that teaches mind-body skills including meditation, autogenics and biofeedback, guided imagery, body awareness, genograms, and self-expression through writing and drawings. The first 4 day training consists of lectures and small groups where the mind-body techniques are practiced. The second 4 day training allows participants to lead a mind-body skills group and teach the techniques under supervision.

SUMMARY:
The goal of this study is to learn about how effective a Mind-Body Medicine Training Program is for prisoners. The main questions it aims to answer are:

1. Does the training program increase resilience?
2. Does the training program reduce depression, anxiety, and/or stress?
3. Does the training program increase optimism?
4. Does the training program increase prisoners' belief that they can have better coping skills?
5. Does the training program increase a sense of meaning in life?
6. Does the training program increase a sense of life purpose?

Participants will attend a 2-part mind-body medicine training program (4 days for each part) and will fill out questionnaires before the training, after the training and 6 months after the training. They will also participate in group interviews after the training and 6 months after the training.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for this study will be English-speaking incarcerated individuals at the Indiana Women's Prison and and at the Plainfield Correctional Facility.

Exclusion Criteria:

1. Having any of the following before the study is completed:

1. a sentence that will end,
2. a scheduled change in security level to a minimum-security prison or,
3. a scheduled work release;

Or 2. Having conduct problems and/or emotional or mental instability that prevents safe and effective participation in the mind-body medicine training program

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on Resilience using the Connor-Davidson Resilience Scale (CD-RISC) after the 8 day training and at 6 month follow-up | Baseline, after the 8 day training, and at 6 month follow-up
  The CD-RISC is a validated, self-report instrument assessing resilience over the last month. The CD-RISC consists of 25 questions that are rated on a 5-point scale with higher scores representing greater resilience. Change = After the 8 day training score- Baseline score; Follow-up score - After the 8 day training score; and Follow-up Score - Baseline score

SECONDARY OUTCOMES:
Change from Baseline on Depression, Anxiety, and Stress using the Depression Anxiety and Stress Scale -21 (DASS-21) after the 8 day training and at 6 month follow-up | Baseline, after the 8 day training, and at 6 month follow-up
  The DASS-21 is a validated, self-report instrument assessing the emotional states of depression, anxiety ans stress over the past week. The DASS-21 consists of 7 questions each for depression anxiety and stress are rated on a 4-point scale with higher scores representing higher levels of depression, anxiety, and stress. Change = After the 8 day training scores- Baseline scores; Follow-up scores - After the 8 day training scores; and Follow-up scores - Baseline scores
Change from Baseline on optimism using the Life Orientation Test - Revised (LOT-R) after the 8 day training and at 6 month follow-up | Baseline, after the 8 day training, and 6 month follow-up
  The LOT-R is a validated, self-report instrument assessing optimism. The LOT-R consists of 10 questions that are rated on a 5-point scale. Four of the questions are "filler questions" and are not calculated in the total score. Higher scores represent greater levels of optimism. Change = After the 8 day training score- Baseline score; Follow-up score - After the 8 day training score; and Follow-up score - Baseline score.
Change from Baseline on coping - self efficacy using the Coping Self-Efficacy (CSE) Scale after the 8 day training and 6 month follow-up | Baseline, after the 8 day training, at 6 month follow-up
  The CSE Scale is a validated, self-report instrument assessing coping self-efficacy. The CSE scale consists of 26 questions that are rated on scale from 0 "cannot do at all" to 10 "certain can do". Higher scores represent greater levels of coping self-efficacy. Change = After the 8 day training score- Baseline score; Follow-up score - After the 8 day training score; and Follow-up score - Baseline score.
Change from Baseline on meaning in life using the Meaning in Life Questionnaire (MLQ) after the 8 day training and 6 month follow-up | Baseline, after the 8 day training, and at 6 month follow-up
  The MLQ is a validated, self-report instrument assessing meaning in life. The MLQ consists of 10 questions that are rated on 7- point scale. There are 2 subscales: presence of meaning and search for meaning. Higher scores represent greater levels of these two components of meaning in life. Change = After the 8 day training score- Baseline score; Follow-up score - After the 8 day training score; and Follow-up score - Baseline score.
Change from Baseline on purpose in life using the Life Engagement Test (LET) after the 8 day training and 6 month follow-up. | Baseline, after the 8 day training, and at 6 month follow-up
  The LET is a 6-item scale made up of items that are framed in half positive and half negative directions. These items are then rated using a 5-point scale that ranges from "1 = strongly disagree" to "5 = strongly agree". Higher scores represent a greater sense of life purpose. Change = After the 8 day training score- Baseline score; Follow-up score - After the 8 day training score; and Follow-up score - Baseline score.

OTHER OUTCOMES:
How the Mind-Body Medicine Training has Affected the Participants by using Focus Group Interviews | After the 8 day training and at 6-month follow-up
  Two focus group interviews will be conducted with approximately 10 participants each. Focus group questions will cover topics such as practice of the mind-body techniques, how the training has affected the participant in terms of relationships, how they view their future, and how they are going to used what they have learned.

CONTACTS AND LOCATIONS:
Overall Officials: Julie K Staples, PhD, Principal Investigator — The Center for Mind-Body Medicine
Locations (1):
- Indiana Department of Correction, Indianapolis, Indiana, United States